CLINICAL TRIAL: NCT01256008
Title: Early Identification and Early Warning of Psychological Problems in Breast Cancer Patients, and Intervention Study Using Cognitive Behavioral Therapy on Depression in Breast Cancer Patients
Brief Title: Intervention Study of Depression in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Collaborators: Anhui Medical University (Other); Central South University (Other); Harbin Medical University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Wuhan University (Other)
Responsible Party: Principal Investigator, Jincai He, Study Chair, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009BAI77B06-3
Record Dates: First submitted 2010-12-06; First posted 2010-12-08 (Estimated); Results first posted 2015-04-10 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Breast Cancer; Depression; Anxiety
Keywords: Breast Cancer; Depression; Anxiety; Cognitive-Behavioral Therapy
MeSH Terms: conditions — Breast Neoplasms; Depression; Anxiety Disorders | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- stage 1 Clinical Management (Placebo Comparator): The group will receive clinical management treatment only each session.
  Interventions: Behavioral: Clinical Management
- stage1 CBT (Experimental): The experimental group will receive CBT
  Interventions: Behavioral: CBT
- stage1 Control group (No Intervention): Participants with breast cancer in the control group received standard medical care, but don't receive any other interventions.

INTERVENTIONS:
Behavioral: CBT — The subjects will receive standardized CBT treatment regularly for 9 sessions(once per week in the first month and once half a month in the second and third months), and each session will last for about 60 minutes.The treatment includes three steps:Concept stage (the first and second sessions): establishment of therapeutic relationships with the subjects; Skills acquisition and repeat stage (the third session to the 8th session): clarification of sources of stress, patients' cognitive and behavioral response to stress. Application and complete price segment (the 9th session): return visit to test efficacy of psychological intervention.
  Other Names: cognitive-behavioral intervention; psychological intervention
  Arms: stage1 CBT
Behavioral: Clinical Management — Clinical management is a clear contrast method of psychological therapy, which is a half-structured interview and lasting for 20-25 minutes each session. Clinical management will be assigned to both experimental group and controlled group in the first stage of intervention.
  Following are major elements:
  Talk to the subjects to find their main problems; introduce knowledge and medication knowledge about cancer and depression; subjects reporting use of drugs for cancer and depression and a variety of signs and symptoms of the reaction. Encourage patients to adhere to drug treatment and to comply with this research program; The operation of CBT and clinical management should be conducted by the same person as far as possible.
  Other Names: Placebo of Cognitive-Behavioral therapy
  Arms: stage 1 Clinical Management

SUMMARY:
The purpose of this study is to evaluate the efficacy of cognitive-behavioral therapy on depression and anxiety in breast cancer patients.

DETAILED DESCRIPTION:
Comprehensive intervention on depression and anxiety in breast cancer patients is a 24-week, multicenter, randomized, blinded controlled clinical study, which uses cognitive-behavioral therapy. This study tries to evaluate the efficacy of sequential therapy on breast cancer patients' depression and its improvement on breast cancer patients' life quality, pain and sleeping.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-65 years;
* Pathologically diagnosed breast cancer patients, with the diagnosis from at least 2 comprehensive clinical attending physicians, in line with clinical diagnosis of breast cancer;
* A week after breast cancer surgery;
* With complaints and symptoms of depression or anxiety
* HAMD-17 ≥ 8 points or / and HAMA ≥ 8 points;
* Have some reading comprehension skills (could complete the self-rating scale independently or with others' help);
* Informed consent

Exclusion Criteria:

* Previous diagnosis of mental disorder or Bipolar Disorder; alcohol and drug abusing history;
* Use antidepressants, antipsychotics or accept any form of psychological treatment, or participation in other clinical trials in the last month
* Patients with cardiovascular disease, liver and kidney dysfunction and other serious diseases;
* Hearing, visual or understanding impairment;
* Severe depression, suicidal tendencies;
* Can not or will not comply with clinical treatment programs based on the physicians' judgment

Exit criteria:

* Persons with poor compliance during the trial period;
* Persons whose depression increased during the trial period, has serious suicidal tendencies and requires urgent intervention;
* Persons who are believed have other circumstances and should be suspended by Physicians

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin C He, MD, Study Chair — Wenzhou Medical University
Locations (1):
- Wenzhou Medical University, Wenzhou, Zhejiang, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1 Clinical Management: The group will receive clinical management treatment only each session.
  Clinical Management: Clinical management is a clear contrast method of psychological therapy, which is a half-structured interview and lasting for 20-25 minutes each session. Clinical management will be assigned to both experimental group and controlled group in the first stage of intervention.
  Following are major elements:
  Talk to the subjects to find their main problems; introduce knowledge and medication knowledge about cancer and depression; subjects reporting use of drugs for cancer and depression and a variety of signs and symptoms of the reaction. Encourage patients to adhere to drug treatment and to comply with this research program; The operation of CBT and clinical management should be conducted by the same person as far as possible.
- Stage 1 CBT: The experimental group will receive CBT each session.
  CBT: The subjects will receive standardized CBT treatment regularly for 9 sessions(once per week in the first month and once half a month in the second and third months), and each session will last for about 60 minutes.The treatment includes three steps:Concept stage (the first and second sessions): establishment of therapeutic relationships with the subjects; Skills acquisition and repeat stage (the third session to the 8th session): clarification of sources of stress, patients' cognitive and behavioral response to stress. Application and complete price segment (the 9th session): return visit to test efficacy of psychological intervention.
- Stage 1 Control Group: Participants with breast cancer in the control group received standard medical care, but don't receive any other interventions.
Period: Overall Study
Arm/Group | Stage 1 Clinical Management | Stage 1 CBT | Stage 1 Control Group
Started | 98 | 98 | 196
Completed | 90 | 91 | 175
Not Completed | 8 | 7 | 21
Not completed — Lost to Follow-up | 6 | 4 | 11
Not completed — Withdrawal by Subject | 2 | 3 | 10

BASELINE CHARACTERISTICS:
Groups:
- stage1 CBT: The experimental group each session.
  CBT: The subjects will receive standardized CBT treatment regularly for 9 sessions(once per week in the first month and once half a month in the second and third months), and each session will last for about 60 minutes.The treatment includes three steps:Concept stage (the first and second sessions): establishment of therapeutic relationships with the subjects; Skills acquisition and repeat stage (the third session to the 8th session): clarification of sources of stress, patients' cognitive and behavioral response to stress. Application and complete price segment (the 9th session): return visit to test efficacy of psychological intervention.
- Total: Total of all reporting groups
Arm/Group | Stage 1 Clinical Management | stage1 CBT | stage1 Control Group | Total
Number analyzed (Participants) | 98 | 98 | 196 | 392
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (8.7) | 46.8 (8.9) | 47.1 (8.3) | 47.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 98 | 196 | 392
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (HAMD-17)
Description: 1. The scale(HAMD-17) is used to assessed the depression symptoms of patients.
  2. The scale range is 0-53.Higher value represents a worse outcome.
  3. The scale was assessed at baseline,2 week,4 week,8 week,12 week,16 week,24 week
Time Frame: baseline,2 w,4 w,8 w,12 w,16 w,24 w
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Stage 1 CBT: The experimental group will receive CBT each session.
  CBT and clinical management: The subjects will receive standardized CBT treatment regularly for 9 sessions(once per week in the first month and once half a month in the second and third months), and each session will last for about 60 minutes.The treatment includes three steps:Concept stage (the first and second sessions): establishment of therapeutic relationships with the subjects; Skills acquisition and repeat stage (the third session to the 8th session): clarification of sources of stress, patients' cognitive and behavioral response to stress. Application and complete price segment (the 9th session): return visit to test efficacy of psychological intervention.
Arm/Group | Stage 1 Clinical Management | Stage 1 CBT | Stage 1 Control Group
Number analyzed (Participants) | 98 | 98 | 196
units on a scale
  baseline | 11.52 (3.789) | 13.31 (5.090) | 11.01 (3.844)
  2W | 10.23 (3.207) | 11.72 (4.976) | 10.28 (3.462)
  4W | 9.80 (3.056) | 9.72 (4.835) | 10.24 (3.688)
  8W | 8.71 (3.601) | 7.80 (4.440) | 9.42 (4.175)
  12W | 8.01 (3.200) | 5.71 (3.979) | 8.81 (4.198)
  16W | 7.42 (3.019) | 5.13 (4.108) | 8.26 (4.338)
  24W | 7.01 (3.317) | 4.45 (3.875) | 7.86 (4.410)

2. Secondary Outcome: Visual Analogue Scale (VAS)
Description: 1. The scale is used to assess the pain intensity of patients.
  2. The scale range of VAS is 0-10. Higher score indicates a higher intensity of pain.
  3. The scale was assessed at baseline,4 week,8 week,12 week,24 week
Time Frame: baseline,4 w,8 w,12 w,24 w
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- stage1 CBT: The experimental group will receive CBT each session.
  CBT: The subjects will receive standardized CBT treatment regularly for 9 sessions(once per week in the first month and once half a month in the second and third months), and each session will last for about 60 minutes.The treatment includes three steps:Concept stage (the first and second sessions): establishment of therapeutic relationships with the subjects; Skills acquisition and repeat stage (the third session to the 8th session): clarification of sources of stress, patients' cognitive and behavioral response to stress. Application and complete price segment (the 9th session): return visit to test efficacy of psychological intervention.
Arm/Group | Stage 1 Clinical Management | stage1 CBT | stage1 Control Group
Number analyzed (Participants) | 98 | 98 | 196
units on a scale
  baseline | 3.23 (2.240) | 3.60 (2.171) | 3.31 (1.956)
  4W | 2.39 (1.907) | 2.48 (2.173) | 2.71 (1.806)
  8W | 2.11 (1.845) | 1.89 (1.899) | 2.41 (1.882)
  12W | 1.92 (1.857) | 1.71 (1.703) | 2.23 (2.025)
  24W | 1.71 (1.982) | 1.45 (1.772) | 2.04 (2.094)

3. Primary Outcome: Hamilton Anxiety Scale (HAMA-14)
Description: 1. The scale(HAMA-14) is used to assessed the anxiety symptoms of patients.
  2. The scale range is 0-56.Higher value represents a worse outcome.
  3. The scale was assessed at baseline,2 week,4 week,8 week,12 week,16 week,24 week.
Time Frame: baseline,2 w,4 w,8 w,12 w,16 w,24 w
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stage 1 Clinical Management | Stage 1 CBT | Stage 1 Control Group
Number analyzed (Participants) | 98 | 98 | 196
units on a scale
  baseline | 12.11 (3.188) | 13.38 (4.883) | 11.37 (2.736)
  2W | 10.89 (3.401) | 11.34 (4.433) | 10.63 (3.105)
  4W | 10.34 (3.505) | 9.82 (3.952) | 10.40 (3.663)
  8W | 9.15 (3.709) | 8.26 (4.120) | 9.36 (3.802)
  12W | 8.57 (3.364) | 6.30 (3.518) | 8.81 (4.231)
  16W | 7.90 (3.263) | 5.42 (3.638) | 8.31 (4.348)
  24W | 7.60 (3.305) | 4.99 (3.263) | 7.91 (4.277)

4. Secondary Outcome: Athens Insomnia Scale(AIS)
Description: 1. The scale is used to assess the sleep quality of patients.
  2. The scale range of AIS is 0-21. Higher score indicates worse sleep quality.
  3. The scale was assessed at baseline,4 week,8 week,12 week,24 week
Time Frame: baseline, 4w,8w,12w,24w
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stage 1 Clinical Management | stage1 CBT | stage1 Control Group
Number analyzed (Participants) | 98 | 98 | 196
units on a scale
  baseline | 6.95 (4.337) | 8.49 (4.341) | 7.14 (4.475)
  4W | 6.06 (3.865) | 5.37 (3.268) | 6.19 (4.235)
  8W | 5.87 (4.414) | 4.22 (3.236) | 5.99 (4.507)
  12W | 5.63 (4.335) | 2.90 (2.242) | 5.85 (4.749)
  24W | 5.34 (4.505) | 2.40 (2.054) | 5.63 (4.946)

5. Secondary Outcome: Functional Assessment of Cancer Treatment (FACT-B)
Description: 1. The scale is used to assess the life quality of patients.
  2. The scale includes 5 subscales. The scores of each scale are summed to compute a total score.
  3. The scale range is 0-144. Higher score indicates better life quality.
  4. The scale was assessed at baseline,4 week,12 week,24 week.
Time Frame: baseline, 4w,12w,24w
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stage 1 Clinical Management | stage1 CBT | stage1 Control Group
Number analyzed (Participants) | 98 | 98 | 196
units on a scale
  baseline | 78.09 (18.86) | 76.78 (19.91) | 79.49 (21.06)
  4W | 80.41 (19.14) | 86.67 (18.74) | 80.07 (22.04)
  12W | 89.69 (16.22) | 102.94 (20.24) | 85.14 (24.61)
  24W | 95.06 (17.54) | 109.21 (19.62) | 89.70 (25.76)

ADVERSE EVENTS:
Groups:
- stage1 CBT: The experimental group will receive CBT each session.
  CBT and clinical management: The subjects will receive standardized CBT treatment regularly for 9 sessions(once per week in the first month and once half a month in the second and third months), and each session will last for about 60 minutes.The treatment includes three steps:Concept stage (the first and second sessions): establishment of therapeutic relationships with the subjects; Skills acquisition and repeat stage (the third session to the 8th session): clarification of sources of stress, patients' cognitive and behavioral response to stress. Application and complete price segment (the 9th session): return visit to test efficacy of psychological intervention.
Arm/Group | Stage 1 Clinical Management | stage1 CBT | stage1 Control Group
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/98 | 0/196
Other Adverse Events (participants affected / at risk) | 0/98 | 0/98 | 0/196

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes